CLINICAL TRIAL: NCT04220125
Title: Preoperative Ketamine as a Strategy to Decrease Perioperative Depression During the Perioperative Period: a Randomized Active Controlled Pilot Study
Brief Title: Preoperative Ketamine and Perioperative Depression
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: No enrollment
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Charles W Hogue, Chair, Department of Anesthesiology, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: STU00211219
Record Dates: First submitted 2020-01-03; First posted 2020-01-07 (Actual); Last update posted 2023-02-06 (Actual); Status verified 2023-02

CONDITIONS: Depressive Disorder
MeSH Terms: conditions — Depressive Disorder | interventions — Ketamine; Midazolam

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Ketamine Group (Experimental): Ketamine 0.5 mg/kg over 40 min via intravenous catheter.
  Interventions: Drug: Ketamine Group
- MIdazolam Group (Active Comparator): Midazolam 0.045 mg/kg administered via intravenous catheter.
  Interventions: Drug: Midazolam injection

INTERVENTIONS:
Drug: Ketamine Group — Ketamine intravenous administration 0.5 mg/kg over 40 minutes.
  Other Names: Ketamine
  Arms: Ketamine Group
Drug: Midazolam injection — Midazolam intravenous administration 0.045 mg/kg IV over 40 minutes.
  Other Names: Midazolam
  Arms: MIdazolam Group

SUMMARY:
Depressive symptoms, in patients with a life history of major depressive disorder (MDD), are very common in the general population, and are especially so in elderly adults undergoing surgery.Symptoms of depression at the time of surgery is associated with risk for postoperative complications.Attenuating depressive symptoms in patients undergoing surgery is thus a plausible but not adequately tested strategy for improving patient postoperative outcomes. Conventional treatment of depression takes weeks and, therefore, is not always a realistic option, particularly when surgery is urgent. Importantly, there are currently no guidelines for diagnosing and managing MDD in surgical patients. Given its association with complications including perioperative cognitive disorders such as delirium, and over longer periods of time with dementing disorders, the feasibility and efficacy of quick-acting treatments for depressive symptoms in surgical patients are direly needed. This need is particularly acute given the rising number of elderly patients undergoing surgery who are prone to depression and surgical complications.

Aim 1: To assess the feasibility of enrolling patients in a clinical trial where a sub-anesthetic dose of ketamine (0.5 mg/kg over 40 min) or midazolam (0.045 mg/kg) is given 1 to 3 days before surgery in the preoperative clinic as a strategy to improve depressive symptoms during the perioperative period.

Aim 2: To obtain estimates of the variability in improvements of depressive symptoms (increase from baseline in MADRS score ≥ 2)1 day after surgery for patients given a sub-anesthetic dose of ketamine (0.5 mg/kg over 40 min) 1 to 3 days before surgery compared with midazolam 0.045 mg/kg.

Aim 3: To assess for the safety and tolerability of administration of a sub-anesthetic dose of ketamine (0.5 mg/kg over 40 min) given 1 to 3 days before surgery in the preoperative clinic (as an outpatient) by assessment of dysphoric symptoms or other complications including the need for hospitalization.

Hypothesis:

Aim 1: Hypothesis: Patients with preoperative depressive symptoms can be identified before surgery and successfully enrolled in a clinical trial comparing a sub-anesthetic dose of ketamine versus midazolam for improving perioperative depressive symptoms.

Aim 2: Hypothesis: Compared with midazolam, a sub-anesthetic dose of ketamine given preoperatively leads to an improvement in MADRS score ≥ 2 on day 1 after surgery.

Aim 3: Hypothesis: Compared with midazolam, a sub-anesthetic dose of ketamine is not associated with dysphoria or other complications.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients age ≥ 65 years
* Planned lumbar surgery for degenerative disc disease or spinal stenosis involving 2 or more levels
* A life history of MDD (DSM-5 criteria) and a MADRS score ≥20
* Mini-Mental State Examination (MMSE) score ≥ 15
* MMSE is between15-26
* Ability to understand English.

Exclusion Criteria:

* MMSE < 15
* History of psychosis
* Poorly controlled hypertension
* Pre-existing aneurysmal vascular disorders
* Cocaine or other illicit drug use.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2023-02-02 (Actual); Study Completion 2023-02-02 (Actual)

PRIMARY OUTCOMES:
Change in depressive symptoms in the perioperative period. | 3 Days before surgery to 30 days after the surgical procedure
  Ketamine administration changes depressive symptoms perioperatively. Measured using Depression will be measured with the Montgomery-Asberg Depression Scale (MADRS) scale. Scale ranges from 0 no depresson- 60 severe depression.

SECONDARY OUTCOMES:
Change in depressive symptoms 1 day after surgery | 24 hours after surgical procedure
  Change in depressive symptoms using MADRS questionnaire measured with the Montgomery-Asberg Depression Scale scale. Scale ranges from 0 no depresson- 60 severe depression.
Safety analsysis of administration of a sub-anesthetic dose of ketamine: CADSS | 65 minutes after study drug has been infused.
  To assess for the safety of administration of a sub-anesthetic dose of ketamine (0.5 mg/kg over 40 min) given 1 to 3 days before surgery in the preoperative clinic (as an outpatient) by assessment of dysphoric symptoms or other complications including the need for hospitalization. The Clinician-Administered Dissociative States Scale CADSS is a 27 question survey ,19 which are completed by the subject on a scale of 0 -4 likert scale for a possible score 0- good 76 poor and 9 questions completed by the assessor (scored yes or no).

CONTACTS AND LOCATIONS:
Overall Officials: Charles Hogue, MD, Principal Investigator — Northwestern University

IPD SHARING:
Plan to Share IPD: No